CLINICAL TRIAL: NCT03881904
Title: Oral Contraceptive Pill Pretreatment in Polycystic Ovary Syndrome Patients Undergoing IVF/ICSI Using the Gonadotrophin Releasing Hormone Antagonist Protocol (A Randomized Controlled Trial)
Brief Title: OCP Pretreatment in PCOS Patients Undergoing ICSI Using Antagonist Protocol
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Khaled Afifi, Assistant lecturer of O&G, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCP-AntagonistPCOS
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Subfertility, Female
Keywords: PCOS; Anatgonist protocol; OCP pretreatment
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCP Group (Active Comparator): This group will include 373 women with PCOS undergoing a trial of IVF/ICSI. This group will receive 0.075mg gestodene/0.03mg ethinylestradiol (Gynera®, Bayer Schering Pharma AG, Germany) from day 2 of the preceding cycle for 21 days followed by GnRH antagonist COH.
  Interventions: Drug: 0.075mg gestodene/0.03mg ethinylestradiol
- Control Group (No Intervention): This group will include 373 women with PCOS undergoing a trial of IVF/ICSI. This group will start GnRH antagonist COH directly without OCP pretreatment.

INTERVENTIONS:
Drug: 0.075mg gestodene/0.03mg ethinylestradiol — OCPs will be started from day 2 of the cycle preceding COH and continued for 21 days, then induction of ovulation using antagonist protocol will be started.
  Other Names: Gynera®
  Arms: OCP Group

SUMMARY:
373 women with PCOS undergoing a trial of IVF/ICSI will receive OCP from day 2 of the preceding cycle for 21 days followed by GnRH antagonist COH.

Another 373 women with PCOS undergoing a trial of IVF/ICSI will start GnRH antagonist COH directly without OCP pretreatment.

Both groups will be followed up for effect on ongoing pregnancy rate.

DETAILED DESCRIPTION:
The study will include 740 women with polycystic ovary syndrome undergoing IVF/ICSI cycle using flexible antagonist protocol.

Randomization:

Patients fulfilling the inclusion criteria will be randomized to two groups.

Study Group:

This group will include 373 women with PCOS undergoing a trial of IVF/ICSI. This group will receive OCP from day 2 of the preceding cycle for 21 days followed by GnRH antagonist COH.

Control Group:

This group will include 373 women with PCOS undergoing a trial of IVF/ICSI. This group will start GnRH antagonist COH directly without OCP pretreatment.

Random allocation sequence generation:

A computer generated list via MedCalc ® Software, version 13.2.2 will be used, assigning each participant number to either study groups.

Allocation Concealment:

Assignment will be done by sequentially numbered, otherwise identical, sealed envelopes (SNOSE), each containing a 2-inch by 2-inch paper with a written code designating the assigned group. These papers will be placed in a folded sheet of aluminum foil fitted inside the envelope. Effort will be taken to assure absence of any detectable differences in size or weight between intervention and control envelopes. Envelopes will be chosen to be opaque and lined inside with carbon paper. Envelopes will be opened sequentially only after writing the subject's tracking information on the envelope so that the carbon paper served as an audit trail.

IVF/ICSI cycle will be done using flexible anatgonist protocol in both groups.

Primary outcome will be ongoing pregnancy rate.

Secondary outcomes will be biochemical and clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-39 years of age.
2. BMI 18-29 Kg/m2
3. Polycystic ovary syndrome, diagnosed - according to the revised 2003 consensus on diagnostic criteria of polycystic ovary syndrome by the Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group - by the presence of two of the following three diagnostic features:

   1. Oligo- or anovulation [defined as fewer than eight episodes of menstrual bleeding per year or menses that occur at intervals greater than 35 days].
   2. Clinical hyperandrogenism [defined by the presence of hirsutism (assessed by a modified Ferriman-Gallwey score ≥ 8), acne or androgenic alopecia] and/or biochemical signs of hyperandrogenism [defined by elevated free androgen index]
   3. Polycystic ovaries [defined as presence of 12 or more follicles in each ovary measuring 2 - 9 mm in diameter, and/or increased ovarian volume > 10 mL) in the early follicular phase (cycle days 3 - 5) in regularly menstruating women. Oligo-/amenorrhoeic women should be scanned either at random or between days 3 and 5 after a progestin-induced withdrawal bleeding. This definition does not apply to women taking oral contraceptive pills, since their use modifies ovarian morphology in normal women and putatively in women with PCO.

   After exclusion of other etiologies (congenital adrenal hyperplasia, androgen secreting tumors, Cushing's syndrome, hypothyroidism and hyperprolactinemia).
4. Normal transvaginal ultrasonography apart from polycystic ovaries (see before).
5. Normal office hysteroscopy.
6. Normal hysterosalpingography.
7. Absence of any structural pathological findings in laparoscopy apart from enlarged sclerotic polycystic ovaries.
8. Normal hormonal profile (apart from hormonal abnormalities associated with PCOS), e.g. normal thyroid function tests
9. Normal parameters of male semen analysis according to WHO criteria 2010.
10. First trial IVF/ICSI.
11. Written and signed informed consent by the patient to participate in the study.

Exclusion Criteria:

1. Age more than 39 years.
2. BMI more than 29 Kg/m2
3. Abnormal ultrasonographic finding, e.g. endometrial polyps, fibroids or ovarian cysts.
4. Abnormal hysteroscopic finding, e.g. endometrial polyps, endometrial hyperplasia or fibroid.
5. Abnormal hysterosalpingographic finding, e.g. hydrosalpinx or peritoneal adhesions.
6. Abnormal male or female karyotyping.
7. Abnormal endocrinological profile during ovarian stimulation not attributed to PCOS, e.g. hypothyroidism, FSH > 12 mIU/mL on day 3.
8. Previous trials of IVF/ICSI.
9. Positive anticardiolipin antibodies or lupus anticoagulant.
10. Positive thrombophilia screen.
11. Abnormal semen analysis parameters according to WHO criteria 2010.
12. Any hormonal treatment within the last 3 months.
13. Any treatment for insulin resistance within the last 3 months, e.g. metformin or leptin.
14. Any chronic medical disorder, e.g. hypertension, autoimmune disorders, … etc.
15. Any category 4 medical condition that contraindicates the usage of OCP according to the WHO Medical eligibility criteria, 2015:

    * Smoking with age ≥ 35 years and cigarettes ≥ 15 /day.
    * Hypertension (systolic ≥ 160 mmHg or diastolic ≥ 90 mmHg).
    * Hypertension with vascular disease.
    * Previous history or acute DVT/PE.
    * Any known thrombogenic mutations.
    * Complicated valvular heart disease.
    * Systemic lupus erythematosus with positive or unkown antiphospholipid antibodies.
    * Migraine with aura.
    * Diabetes with nephropathy/neuropathy/retinopathy.
    * Diabetes > 20 years.
    * Acute hepatitis, severe cirrhosis or liver tumors.
16. Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 740 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 20 gestational weeks
  Number of pregnancies completing ≥20 weeks gestational age expressed per 100 embryo transfer cycles

SECONDARY OUTCOMES:
Chemical pregnancy rate | 6 gestational weeks
  Number of biochemical pregnancies (evidenced by positive pregnancy test in serum or urine without ultrasound evidence of a gestational sac) expressed per 100 embryo transfer cycles
Clinical pregnancy rate | 6 gestational weeks
  Number of clinical pregnancies (evidenced by ultrasound visualization of a gestational sac and embryonic pole with heartbeat) expressed per 100 embryo transfer cycles
Live birth rate | 38 gestational weeks
  The number of deliveries (> 28 weeks GA) that resulted in a live born neonate, expressed per 100 embryo transfers

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Fouad, MD, Principal Investigator — Assistant Professor; Ahmed Abbas, MD, Study Director — Lecturer
Locations (1):
- AinShams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No